CLINICAL TRIAL: NCT04653610
Title: Sequential Analysis Before and After Treatment Initiation to Unravel the Role of Naturally Occurring Extracellular Vesicles in HIV Infection
Acronym: Saturne-HIV
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: BC-08408
Record Dates: First submitted 2020-10-23; First posted 2020-12-04 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Hiv
Keywords: HIV; Extracellular Vesicles
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HIV-infected individuals
- HIV-seronegative healthy volunteers

SUMMARY:
This study aims to evaluate the role of extracellular vesicles in HIV-infection, by determining the expression profile and content of EVs before and after treatment initiation in HIV-infected patients, through extensive blood and tissue sampling (leukapheresis, stool sampling and colon biopsies). A one-time sampling (blood, stool, colon biopsies) will also be performed in HIV-seronegative healthy volunteers to confirm that results found in HIV-infected patients are related to the disease.

ELIGIBILITY:
A. HIV-infected individuals

A.1. Inclusion Criteria:

* Documented untreated HIV-1 infection defined as followed: HIV-1-specific antibody+(western blot); p31+ (ELISA)
* CD4 T cell count will be determined standard of care (SOC). A minimum of 16 patients will be included with a CD4 T cell count lower than 350 cells/µl and a minimum of 16 patients with a CD4 T cell count higher than 350 cells/µl
* Able and willing to provide written informed consent
* Age ≥ 18 years and ≤ 65 years
* Ability to attend the complete schedule of assessments and patient visits as described in the schedule below
* Ability and willingness to have blood, stool and colon samples collected and stored for 20 years after finalizing the study, and used for various research purposes

A.2. Exclusion Criteria:

* Recent HIV-infection, early diagnosis
* Previous or current history of opportunistic infection (AIDS defining events as defined in category C of the CDC clinical classification), consisting of chronic HIV-1 infection
* Evidence of active HBV infection (Hepatitis B surface antigen positive or HBV viral load positive in the past and no evidence of subsequent seroconversion (=HBV antigen or viral load negative and positive HBV surface antibody))
* Evidence of active HCV infection: HCV antibody positive result within 60 days prior to study entry with positive HCV viral load or, if the HCV antibody result is negative, a positive HCV RNA result within 60 days prior to study entry
* Current or known history of cardiomyopathy or significant ischemic or cerebrovascular disease
* Current or known history of cancer
* Pregnancy or breastfeeding
* Any conditions, including preexisting psychiatric and psychological disorders, which will in the opinion of the investigator interfere with the trial conduct or safety of the participant. An initial psychiatric assessment will be made by the treating physician. Since making a correct psychological assessment at the time of diagnosis can be difficult, a visit with a psychologist is planned for patients included in the study, for a second evaluation. This will be planned within the first month after diagnosis. In consultation with the psychologist, further sampling will be planned or the patient will be excluded from further sampling.
* Previous participation in a trial evaluating an immune modulating agent
* Abnormal laboratory tests results at screening:

  1. Confirmed hemoglobin <11g/dl for women and <12 g/dl for men
  2. Confirmed platelet count < 100 000/µl
  3. Confirmed neutrophil count <1000/μl
  4. Confirmed AST and/or ALT > 10x ULN
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements
* Acute or serious illness, in the opinion of the site investigator, requiring systemic treatment and/or hospitalization within 60 days prior to entry
* Known inflammatory bowel disease (Crohn's disease or ulcerative colitis)

B. Healthy Volunteers

B.1. Inclusion Criteria:

* Able and willing to provide written informed consent
* Age ≥ 18 years and ≤ 65 years
* Ability to attend the complete sampling schedule, as described below
* Ability and willingness to have blood, stool and colon samples collected and stored for 20 years and used for various research purposes

B.2. Exclusion Criteria:

* HIV-infection
* Evidence of active HBV infection (Hepatitis B surface antigen positive or HBV viral load positive in the past and no evidence of subsequent seroconversion (=HBV antigen or viral load negative and positive HBV surface antibody))
* Evidence of active HCV infection: HCV antibody positive result within 60 days prior to study entry with positive HCV viral load or, if the HCV antibody result is negative, a positive HCV RNA result within 60 days prior to study entry
* Current or known history of cardiomyopathy or significant ischemic or cerebrovascular disease
* Current or known history of cancer
* Pregnancy or breastfeeding
* Any conditions, including preexisting psychiatric and psychological disorders, which will in the opinion of the investigator interfere with the trial conduct or safety of the participant
* Previous participation in a trial evaluating an immune modulating agent
* Abnormal laboratory tests results at screening:

  1. Confirmed hemoglobin <11g/dl for women and <12 g/dl for men
  2. Confirmed platelet count < 100 000/µl
  3. Confirmed neutrophil count <1000/μl
  4. Confirmed AST and/or ALT > 10xULN
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements
* Acute or serious illness, in the opinion of the site investigator, requiring systemic treatment and/or hospitalization within 60 days prior to entry
* Known inflammatory bowel disease (Crohn's disease or ulcerative colitis)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Our aim is to enroll a minimum of 32 and a maximum of 50 untreated HIV-infected patients. We aim to include a minimum of 16 patients with a CD4 T cell count lower than 350 cells/µl and a minimum of 16 patients with a CD4 T cell count higher than 350 cells/µl. Of the HIV-infected patients, we aim to include 12 patients undergoing additional sampling consisting of lymph node excisions and an ileocolonoscopy (see below).
  Furthermore we aim to include 55 HIV-negative "healthy donors", from which we will collect inguinal lymph node samples, gut biopsies, a blood draw or leukapheresis and stool sample to confirm that the results found in HIV-patients are related to the disease. HIV seronegative participants can choose which procedures they would like to undergo, it is not necessary to undergo all study-related procedures. Before sampling, patients and healthy volunteers willing to participate will be enrolled following informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2021-01-27 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Extracellular Vesicles analysis-NTA | 6 years
  Extracellular vesicles (EV) will be isolated through a combination of size-exclusion chromatography (SEC) and Optiprep density gradient (ODG). Nanoparticle Tracking Analysis (NTA) will be performed to obtain the concentration and size distribution of EVs in the samples.
Extracellular Vesicles analysis-microscopy | 6 years
  The isolated EVs will be further visualized by (electron) microscopy.
Extracellular Vesicles analysis-western blot | 6 years
  The isolated EVs will be further characterized through western blot.
Extracellular Vesicles analysis-PCR | 6 years
  The isolated EVs will be further characterized through PCR.
Extracellular Vesicles analysis-proteomics | 6 years
  The isolated EVs will be further characterized through proteomic analysis.
Extracellular Vesicles analysis-RNAsequencing | 6 years
  The isolated EVs will be further characterized through RNA sequencing.
Extracellular Vesicles analysis-reporter assays | 6 years
  Reporter assays will be performed to quantitatively measure bacterial EV-associated lipopolysaccharide (LPS).
Quantification of HIV DNA and RNA | 6 years
  Digital PCR
Immunological analysis-FACS | 6 years
  Immunophenotyping by flow cytometric assays will be performed of different cells to assess the phenotype of innate immune cells, using FACS analysis.
Immunological analysis-ELISA | 6 years
  Immunophenotyping by flow cytometric assays will be performed of different cells to assess the phenotype of innate immune cells, using ELISA.
Gene expression analysis/transcriptomics | 6 years
Microbiome monitoring | 6 years
  Gut microbiome will be analyzed in stool and colon biopsies using next-generation sequencing (NGS) of rRNA gene amplicons to identify bacteria at genus/species level
Virological analysis-FLIPS | 6 years
  HIV will be characterized by Full Length Individual Proviral Sequencing (FLIPS).
Virological analysis-integration site | 6 years
  HIV will be characterized by integration site analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Linos Vandekerckhove, Prof. Dr., Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: Undecided